CLINICAL TRIAL: NCT04050462
Title: A Phase II, Randomized, Controlled Trial of Nivolumab in Combination With BMS-986253 in Advanced Hepatocellular Carcinoma (HCC) Patients
Brief Title: Nivolumab Combined With BMS-986253 in HCC Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early by the drug sponsor due to slow accrual and a change in the company's drug development priorities
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01028
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; cabiralizumab; HuMax-IL8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab Monotherapy (Active Comparator)
  Interventions: Drug: Nivolumab 240 mg IV every 2 weeks
- Nivolumab/BMS-986253 combination (Experimental)
  Interventions: Drug: Nivolumab 240 mg IV every 2 weeks + BMS-986253 1200 mg IV every 2 weeks; Drug: Nivolumab 240 mg IV every 2 weeks
- Nivolumab/Cabiralizumab combination (Experimental)
  Interventions: Drug: Nivolumab 240 mg IV every 2 weeks + Cabiralizumab 4 mg/kg IV every 2 weeks; Drug: Nivolumab 240 mg IV every 2 weeks

INTERVENTIONS:
Drug: Nivolumab 240 mg IV every 2 weeks + Cabiralizumab 4 mg/kg IV every 2 weeks — Nivolumab 240 mg IV plus Cabiralizumab 4 mg/kg IV every 2 weeks combination therapy
  Arms: Nivolumab/Cabiralizumab combination
Drug: Nivolumab 240 mg IV every 2 weeks + BMS-986253 1200 mg IV every 2 weeks — Nivolumab 240 mg IV plus BMS-986253 1200mg IV every 2 weeks
  Arms: Nivolumab/BMS-986253 combination
Drug: Nivolumab 240 mg IV every 2 weeks — Arm 1 (control) Nivolumab 240mg IV every 2 weeks monotherapy

SUMMARY:
A phase II clinical trial is utilized to examine whether BMS-986253 (25 subjects) or Cabiralizumab (25 subjects) when combined with Nivolumab offers improved radiographic objective response rates (ORR) over Nivolumab monotherapy (25 subjects) in advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed evidence of HCC, Childs-Pugh score of ≤7.

   a. Participants must be willing to provide specimen from fresh, pre- and on-treatment tumor core biopsies for histologic diagnosis and translational studies.
2. Radiographically measurable disease by RECIST1.1 in at least one site.
3. Deemed to not be a candidate for resection or other local-regional therapy.
4. Must not be receiving treatment with other investigational agents and must not have received any other systemic therapy prior to registration.

   a. Prior radioembolization, local ablative therapies (radiofrequency, microwave or cryoablation), radiation (external beam or stereotactic), or hepatic resection permitted if completed ≥ 4 weeks prior to study enrollment and if patient has recovered with ≤ grade 1 toxicity and if untreated measurable disease is present.
5. Be willing and able to provide written informed consent/assent for the trial.
6. Participants must be ≥ 18 years
7. Have a Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
8. If hepatitis B is present, participants must be on anti-viral HBV therapy.
9. All women of childbearing potential (not surgically sterilized and between menarche and 1 year post menopause) must have a blood test to rule out pregnancy within 24 hours prior to start of study treatment
10. All women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment (s) and for 5 months following discontinuation of study treatment.
11. Males who are sexually active with women of childbearing potential must agree to follow instructions for method (s) of contraception for the duration of treatment with study treatment and for 7 months following discontinuation of study treatment. Additionally, male participants must not donate sperm during this period.
12. Demonstrate adequate organ function as defined by the following required lab and acceptable range criteria:

Adequate bone marrow function:

Absolute neutrophil count > 1000/mcL Platelet count > 50,000/mcL Hemoglobin > 8.5 g/dL

Adequate hepatic function:

Total bilirubin < 2 mg/dL or < 1.5 times upper limit of normal (ULN) AST and ALT < 5 times ULN INR < 1.5 times ULN Albumin > 2.8 g/dL

Adequate renal function:

Creatinine < 2.0 mg/Dl

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Presence of other malignancies. Participants with active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ. NOTE: Patients with history of malignancy are not considered to have a "currently active" malignancy if they have completed therapy and are now considered by their physician to be at less than 30% risk for relapse.
3. Have active or history of Tuberculosis
4. Participants with known HIV positive status
5. Participants with known CNS metastases
6. Uncontrolled ascites
7. Uncontrolled encephalopathy
8. Uncontrolled gastro-esophageal varicesPrior organ allograft or allogeneic bone marrow transplantation
9. Participants with active, known, or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study treatment), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
10. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study treatment administration except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease. Note: Treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study treatment is permitted.
11. Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity.
12. Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

    * Myocardial infarction or stroke/transient ischemic attack within the past 6 months
    * Uncontrolled angina within the past 3 months
    * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
    * History of other clinically significant heart disease (eg, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, significant pericardial effusion, or myocarditis)
    * Cardiovascular disease-related requirement for daily supplemental oxygen therapy.
13. Participants with ongoing or active, uncontrolled infections (afebrile for ≥ 48 hours off antibiotics). If hepatitis B is present, must be on anti-viral HBV therapy.
14. Must not have a psychiatric illness, other significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements.
15. Any major surgery within 4 weeks of study treatment. Participants must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before
16. Any uncontrolled inflammatory disease including Crohn's disease and ulcerative colitis
17. Treatment with botanical preparations (eg, herbal supplements, including potential drugs of abuse, or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to randomization/treatment.
18. Concomitant use of statins while on study.
19. Current or history of clinically significant muscle disorders (eg, myositis), recent unresolved muscle injury, or any condition known to elevate serum CK levels.
20. Known history of sensitivity to infusions containing Tween 20 (polysorbate 20) and Tween 80 (polysorbate 80).
21. Participants who have received a live / attenuated vaccine within 30 days of first treatment.
22. Concomitant use of any live / attenuated vaccine during treatment and until 100 days following last dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Beri, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab Monotherapy | Nivolumab/BMS-986253 Combination | Nivolumab/Cabiralizumab Combination
Started | 6 | 7 | 0
Completed | 5 | 7 | 0
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were included in the baseline data analysis. The data were analyzed based on intention-to-treat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab Monotherapy | Nivolumab/BMS-986253 Combination | Nivolumab/Cabiralizumab Combination | Total
Number analyzed (Participants) | 6 | 7 | 0 | 13
Age, Continuous [Median (Full Range); unit: years] | 72.5 [62 to 77] | 70 [48 to 77] |  | 70 [48 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 |  | 2
  Male | 5 | 6 |  | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 |  | 2
  Not Hispanic or Latino | 6 | 5 |  | 11
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 2 | 2 |  | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 1 | 0 |  | 1
  White | 3 | 4 |  | 7
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 |  | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is measured as the percentage of people in a study or treatment group who have a partial response or complete response to the treatment. ORR will be determined based upon RECIST v. 1.1 criteria. Per RECIST v. 1.1 criteria, a Complete Response (CR) is the disappearance of all target lesions, and a Partial Response (PR) is at least a 30% decrease in the sum of the longest diameters (LD) of the target lesions, compared to the baseline.
Time Frame: Every 8 weeks for 1 year and every 3 months thereafter (assessed up to 5 years)
Population: 1 subject on the monotherapy arm withdrew consent after randomization, prior to starting treatment
Measure: Number; unit: percentage of particpants
Arm/Group | Nivolumab Monotherapy | Nivolumab/BMS-986253 Combination | Nivolumab/Cabiralizumab Combination
Number analyzed (Participants) | 5 | 7 | 0
percentage of particpants | 20 | 28.57 |

2. Secondary Outcome: Time to Response (TTR)
Description: TTR is the amount of time it takes for a tumor to show a measurable decrease in size or other signs of response after treatment begins
Time Frame: From treatment initiation until first sign of response (up to 5 years)
Population: Number of subjects who showed response in each arm were included in analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Nivolumab Monotherapy | Nivolumab/BMS-986253 Combination | Nivolumab/Cabiralizumab Combination
Number analyzed (Participants) | 1 | 2 | 0
days | 126 [126 to 126] | 116 [115 to 117] |

3. Secondary Outcome: Disease Control Rate (DOR)
Description: DOR is the percentage of patients who experience either a complete response (CR), a partial response (PR), or stable disease (SD) to a treatment
Time Frame: Through study completion (assessed up to 5 years)
Population: 1 subject on the monotherapy arm withdrew consent after randomization, prior to starting treatment
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab Monotherapy | Nivolumab/BMS-986253 Combination | Nivolumab/Cabiralizumab Combination
Number analyzed (Participants) | 5 | 7 | 0
percentage of participants | 80 | 57.14 |

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is measured as the time from the date of enrollment to disease progression per RECIST v. 1.1 criteria.
Time Frame: From date of treatment until the date of first documented progression (assessed up to 5 years)
Population: 1 subject on the monotherapy arm withdrew consent after randomization, prior to starting treatment
Measure: Median (Full Range); unit: days
Arm/Group | Nivolumab Monotherapy | Nivolumab/BMS-986253 Combination | Nivolumab/Cabiralizumab Combination
Number analyzed (Participants) | 5 | 7 | 0
days | 191 [57 to 1995] | 171 [52 to 985] |

5. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from treatment start to death of participants.
Time Frame: From date of treatment until the date of death from any cause (assessed up to 5 years)
Population: 1 subject on the monotherapy arm withdrew consent after randomization, prior to starting treatment
Measure: Median (Full Range); unit: days
Arm/Group | Nivolumab Monotherapy | Nivolumab/BMS-986253 Combination | Nivolumab/Cabiralizumab Combination
Number analyzed (Participants) | 5 | 7 | 0
days | 465 [145 to 1995] | 409 [127 to 1422] |

ADVERSE EVENTS:
Time Frame: AEs and SAEs are assessed from the time of consent until 100 days following the last administration of study treatment (through study completion, up to 64 months)
Description: Treating physicians assess AEs at every office visit; participants are encouraged to call the research team and self-report any AEs in-between visits.
Arm/Group | Nivolumab Monotherapy | Nivolumab/BMS-986253 Combination | Nivolumab/Cabiralizumab Combination
All-Cause Mortality (participants affected / at risk) | 0/6 | 2/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/7 | 0/0
Other Adverse Events (participants affected / at risk) | 5/6 | 7/7 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Monotherapy (N=6) | Nivolumab/BMS-986253 Combination (N=7) | Nivolumab/Cabiralizumab Combination (N=0)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Fever (General disorders) | 0 | 1 | 0
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Peripheral Ischemia (Vascular disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin Infection (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Thromboembolic Event (Vascular disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Monotherapy (N=6) | Nivolumab/BMS-986253 Combination (N=7) | Nivolumab/Cabiralizumab Combination (N=0)
Abdominal Pain (Gastrointestinal disorders) | 2 | 4 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 3 | 0
Alkaline Phosphatase Increased (Investigations) | 1 | 5 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 5 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 3 | 4 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Bloating (Gastrointestinal disorders) | 1 | 1 | 0
Blood And Lymphatic System Disorders (Blood and lymphatic system disorders) | 0 | 2 | 0
Blood Bilirubin Increased (Investigations) | 1 | 3 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest Pain (Cardiac disorders) | 0 | 2 | 0
Chills (General disorders) | 1 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Creatinine Increased (Investigations) | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Edema Limbs (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Enterocolitis Infectious (Infections and infestations) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Eye Disorders (Eye disorders) | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 0
Fatigue (General disorders) | 3 | 3 | 0
Fever (General disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Flu Like Symptoms (General disorders) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 | 1 | 0
General Disorders And Administration Site Conditions (General disorders) | 1 | 2 | 0
Headache (Vascular disorders) | 1 | 3 | 0
Hematoma (Vascular disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 6 | 0
Infections And Infestations (Infections and infestations) | 1 | 1 | 0
INR Increased (Investigations) | 2 | 3 | 0
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0 | 0
Investigations (Investigations) | 0 | 1 | 0
Lipase Increased (Investigations) | 0 | 1 | 0
Localized Edema (General disorders) | 0 | 1 | 0
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 5 | 0
Lymphocyte Count Increased (Investigations) | 0 | 1 | 0
Metabolism And Nutrition Disorders (Metabolism and nutrition disorders) | 0 | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 1 | 1 | 0
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal And Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nail Changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 2 | 0
Pain (General disorders) | 3 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 3 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rash Maculo (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Serum Amylase Increased (Investigations) | 0 | 1 | 0
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin Infection (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Weight Gain (Investigations) | 0 | 1 | 0
Weight Loss (Investigations) | 0 | 1 | 0
White Blood Cell Decreased (Investigations) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT04050462/Prot_SAP_000.pdf